CLINICAL TRIAL: NCT04436952
Title: An Open Label Study to Compare and Evaluate the Efficacy of the Deep Transcranial Magnetic Stimulation With and Without Exposure and Response Prevention (ERP) to Repetitive Transcranial Magnetic Stimulation With and Without ERP to ERP.
Brief Title: Is There a New Gold Standard for the Treatment of Obsessive-Compulsive Disorder?
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in Protocol
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENV-OCD-2020-01
Record Dates: First submitted 2020-05-23; First posted 2020-06-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2020-06

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Obsessive Compulsive Disorder; Transcranial Magnetic Stimulation; Exposure and Response Prevention
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: 1. Group 1 - 20 patients undergoing DTMS treatment using the H7 coil
  2. Group 2 - 20 patients undergoing rTMS treatment using the cool D-B80 coil
  3. Group 3 - 20 patients undergoing DTMS treatment using the H7 coil + ERP
  4. Group 4 - 20 patients undergoing rTMS treatment using the cool D-B80 coil + ERP
  5. Group 5 - 20 patients undergoing ERP only
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (5):
- H7 coil only (Experimental): patients undergoing DTMS treatment using the H7 coil
  Interventions: Device: H7 coil
- Cool D-B80 coil only (Active Comparator): 20 patients undergoing rTMS treatment using the cool D-B80 coil
  Interventions: Device: Cool D-B80
- DTMS treatment using the H7 coil + ERP (Active Comparator): 20 patients undergoing DTMS treatment using the H7 coil + ERP
  Interventions: Device: H7 coil; Behavioral: Exposure Response Prevention (ERP)
- rTMS treatment using the cool D-B80 coil + ERP (Active Comparator): 20 patients undergoing rTMS treatment using the cool D-B80 coil + ERP
  Interventions: Device: Cool D-B80; Behavioral: Exposure Response Prevention (ERP)
- ERP only (Active Comparator): 20 patients undergoing ERP only
  Interventions: Behavioral: Exposure Response Prevention (ERP)

INTERVENTIONS:
Device: H7 coil — The H7 coil arm will receive a medial prefrontal cortex (mPFC) DTMS 5 days a week for 8 consecutive weeks = 40 Sessions 20 Hz at 100% MT, 2 s on 20 s off intertrain interval, 50 trains, 2000 stimuli per session.
  Arms: DTMS treatment using the H7 coil + ERP; H7 coil only
Device: Cool D-B80 — The Cool D-B80 arm will receive dorsomedial prefrontal cortex (DMPFC) rTMS 5 days a week for 8 consecutive weeks = 40 sessions 10 Hz at 120% MT, 5 s on 10 s off intertrain interval, 60 trains, First 3000 pulses to the left DMPFC then 3000 pulses to the right DMPFC. TMS will be done at active state by provocation
  Arms: Cool D-B80 coil only; rTMS treatment using the cool D-B80 coil + ERP
Behavioral: Exposure Response Prevention (ERP) — The ERP will be conducted for 2 hours on week 1 and week 8 and for 1 hour on Weeks 2 to 7 for a total of 10 hours
  Arms: DTMS treatment using the H7 coil + ERP; ERP only; rTMS treatment using the cool D-B80 coil + ERP

SUMMARY:
Obsessive Compulsive Disorder is a highly debilitating condition with a lifetime prevalence of 2%-3%, and a notable percentage of patients (40-60%) have a partial or no response to medications. The present gold standard for the treatment of OCD is medications (Selective serotonin reuptake inhibitors (SSRIs) / Clomipramine) + Exposure and Response Prevention (ERP). There is a significant need for alternative novel methods of treatment. One of the novel methods of treating OCD is using magnetic stimulation which has already been successfully used in the treatment of depression. Treating OCD is difficult with regular superficial repetitive Transcranial Magnetic Stimulation (rTMS) hence the need for coils that targets deeper structures. Thus, we are comparing the efficacy of the two different coils from two different manufacturers plus using ERP in combination with the different coils.

1. Deep Transcranial Magnetic Stimulation (DTMS) using BrainsWay H7 coil targets deeper structures such as medial prefrontal cortex. The H7 coil has already shown clear evidence in treating patients with OCD and has been approved by the FDA for clinical use.
2. Repetitive Transcranial Magnetic Stimulation (rTMS) using MagVenture Cool D-B coil could also target the medial prefrontal cortex. Hence it might also be equally effective as the BrainsWay H7 coil in treating patients with OCD.

DETAILED DESCRIPTION:
i. Purpose

a) The purpose of this study is to compare and evaluate the efficacy of repetitive Transcranial Magnetic Stimulation (rTMS) by MagVenture and Deep Transcranial Magnetic Stimulation (DTMS) by BrainsWay with and without the combination of active Exposure and Response Prevention (ERP) for the treatment of patients with OCD.

ii. Hypothesis a) We hypothesize that the combination of TMS + active ERP will have a superior efficacy in the treatment of OCD. We also hypothesize that MagVenture cool D-B80 coil will be as effective as BrainsWay H7 coil in treating patients with OCD.

iii. Justification

1. The Prospective Multicenter Randomized Double-Blind Placebo-Controlled Trial by Carmi et al. (2019) had shown significant improvement in OCD symptoms by using the H7 coil and provocation of OCD symptoms before and during treatment.
2. The study by Dunlop et al. (2016) has shown reduction in OCD symptom severity by using the Cool D-B80 Coil without provocation.
3. There have been no head to head studies comparing the BrainsWay H7 coil and MagVenture Cool D-B80 coil using provocation methods for both coils.
4. Also there have been no head to head studies comparing the gold standard treatment of medications + active ERP with medications + active ERP + TMS and medications + TMS.

iv. Objectives

a) The aim of the study is to evaluate and compare the efficacy of DTMS treatment and the rTMS treatment with and without the combination of active ERP in patients suffering from OCD, in conjunction with medications approved for OCD treatment.

v. Research Method/Procedure

1. Recruit 100 patients suffering from OCD who have been treated and currently on at least one SSRIs, SNRIs, clomipramine and at least one trial of CBT (Exposure and Response Prevention) had an inadequate response.
2. Make a personalized provocation for each patient and using them during treatment
3. The trial will consist of 3 phases:

   1. Pre-study screening and baseline assessment;
   2. Treatment trial period (8 weeks); and
   3. Follow-up (12 weeks).
4. Clinical severity rating scales will be taken every other week and include: (Brief Obsessive-Compulsive Scale (BOCS), Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) , Beck's Depression Inventory (BDI), Clinical Global Impression Severity (CGI-S) and Clinical Global Impression Improvement (CGI-I). Safety evaluations will include adverse event monitoring, vital signs, and cognitive changes (Mini-Mental State Exam (MMSE)). All measures will be taken before treatment administration.
5. Pre-Study Screening and Baseline Assessment

   1. Potential Patients will be given complete information describing the study treatment and their role in the trial, and they will be encouraged to ask any questions regarding the trial. The risks and requirements of this clinical research trial will be explained to each potential patient. Those volunteering to take part will read and sign the Informed Consent Form for participation in the clinical research trial before any trial-related procedures are performed.
   2. Upon obtaining the signed informed consent, inclusion and exclusion criteria will be reviewed to verify the patient's eligibility.
   3. Baseline data are defined as the data generated during the baseline visit before the first treatment Session.
6. After the patients has been admitted into the study, they will be asked to undergo a fMRI and then randomly organized based on age and symptom severity into the 5 different groups.
7. Comparing 5 groups of patients with OCD 1) Group 1 - 20 patients undergoing DTMS treatment using the H7 coil 2) Group 2 - 20 patients undergoing rTMS treatment using the cool D-B80 coil 3) Group 3 - 20 patients undergoing DTMS treatment using the H7 coil + ERP 4) Group 4 - 20 patients undergoing rTMS treatment using the cool D-B80 coil + ERP 5) Group 5 - 20 patients undergoing ERP only
8. Treatment Trial period

   1) During the treatment phase the patients will either receive

   Group 1 - medial prefrontal cortex (mPFC) DTMS 5 days a week for 8 consecutive weeks = 40 Sessions 20 Hz at 100% MT, 2 s on 20 s off intertrain interval, 50 trains, 2000 stimuli per session.

   TMS will be done at active state by provocation

   Group 2 - dorsomedial prefrontal cortex (DMPFC) rTMS 5 days a week for 8 consecutive weeks = 40 sessions 10 Hz at 120% MT, 5 s on 10 s off intertrain interval, 60 trains, First 3000 pulses to the left DMPFC then 3000 pulses to the right DMPFC. TMS will be done at active state by provocation

   Group 3 - medial prefrontal cortex (mPFC) DTMS + ERP 5 days a week for 8 consecutive weeks = 40 sessions 20 Hz at 100% MT, 2 s on 20 s off intertrain interval, 50 trains, 2000 stimuli per session. TMS will be done at active state by provocation The ERP will be administered for 2 hours on week 1 and week 8 and for 1 hour on Weeks 2 to 7 for a total of 10 hours.

   Group 4 - dorsomedial prefrontal cortex (DMPFC) rTMS +ERP 5 days a week for 8 consecutive weeks = 40 sessions 10 Hz at 120% MT, 5 s on 10 s off intertrain interval, 60 trains, First 3000 pulses to the left DMPFC then 3000 pulses to the right DMPFC. TMS will be done at active state by provocation The ERP will be administered for 2 hours on week 1 and week 8 and for 1 hour on Weeks 2 to 7 for a total of 10 hours.

   Group 5 - ERP The ERP will be conducted for 2 hours on week 1 and week 8 and for 1 hour on Weeks 2 to 7 for a total of 10 hours.
9. Prior to initiation and during each treatment of TMS, OCD symptoms will be provoked for each patient in an individual manner to activate the relevant brain circuitry. Targeted questions will be designed for each patient using external, internal or a combination of provocations and the degree of provocation on a Visual Analog Scale will be recorded. These may require adjustment as the patient improves.
10. Study evaluations will be performed every week at the beginning of the next treatment week (from week 2), prior to the first or second (preferably second) treatment session of that week. Procedures to be performed at the 8-week visit will also be performed in case of Early Discontinuation of the study.
11. Follow up period 1) All patients will be followed up at week 12. vi. Plan for Data Analysis

<!-- -->

1. Primary Efficacy Variable

   - The primary outcome measure is the BOCS and YBOCS severity rating scale. The primary efficacy endpoint is the change in BOCS and YBOCS severity score from baseline to the 8-week visit.
2. Secondary Efficacy Variables

   - Change from baseline to the 8-week visit in the Clinical Global Impression - Severity (CGI-S) and Improvement (CGI-I) scores.

   - Change from baseline to the 12-week visit in the BOCS and YBOCS severity score.

   - Change from baseline to the 12-week visit in the Clinical Global Impression - Severity (CGI-S) and Improvement (CGI-I) scores.
3. Exploratory Efficacy Variables - Change from baseline to the 8 week and 12 weeks visit in the Beck's Depression Inventory score.

   * fMRI changes before and after treatment and using fMRI to predict future response to TMS treatment (to identify responders and non-responders)

ELIGIBILITY:
Inclusion Criteria:

i. Outpatients ii. Men and women 18-70 years of age. iii. Patients diagnosed as suffering from OCD according to the BOCS and YBOCs. iv. Patients had an inadequate/intolerable response to SSRI, CBT (Exposure and Response Prevention) or both.

v. Patient is capable and willing to provide informed consent, and their guardians is capable of providing informed consent.

vi. Patient is able to adhere to the treatment schedule.

Exclusion Criteria:

i. Present suicidal risk is significant as assessed during the investigator's mental status exam and psychiatric interview.

ii. Patient has a history of epilepsy or seizure (EXCEPT those therapeutically induced by ECT) or history of such in first-degree relatives.

iii. Patient has an increased risk of seizure for any reason, including prior diagnosis of increased intracranial pressure, or history of significant head trauma with loss of consciousness for greater than or equal to 5 minutes.

iv. Patient has a history of head injury necessitating cranial surgery or prolonged coma.

v. Patient has ferromagnetic material in the head including the eyes and ears (outside the mouth) and body.

vi. Patient has a history of significant hearing loss. vii. Patients with significant neurological disorder or insult including, but not limited to:

1. Any condition likely to be associated with increased intracranial pressure
2. Space occupying brain lesion
3. History of cerebrovascular accident
4. Transient ischemic attack within two years
5. Cerebral aneurysm
6. Dementia
7. Parkinson's disease
8. Huntington's chorea
9. Multiple sclerosis
10. Mini Mental State Exam score of less than or equal to 24 (for adult participants) viii. Patient has a history of substance abuse including alcohol use disorder within the past 6 months (except nicotine and caffeine).

ix. Inadequate communication with the patient. x. Patient is currently participating in another clinical study or enrolled in another clinical study within 30 days prior to this study.

xi. Patients who suffer from an unstable physical, systemic and metabolic disorder such as unstable blood pressure or acute, unstable cardiac disease.

xii. Women who are pregnant or with suspected pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Reduction in the severity of OCD symptoms | 8 weeks
  - The primary outcome measure is the BOCS and YBOCS severity rating scale. The primary efficacy endpoint is the change in BOCS and YBOCS severity score from baseline to the 8-week visit.

SECONDARY OUTCOMES:
Clinical Global Impression - Severity (CGI-S) and Improvement (CGI-I) scores. | 8-12 weeks
  Change from baseline to the 8-week visit in the Clinical Global Impression - Severity (CGI-S) and Improvement (CGI-I) scores.
  Change from baseline to the 12-week visit in the BOCS and YBOCS severity score. Change from baseline to the 12-week visit in the Clinical Global Impression - Severity (CGI-S) and Improvement (CGI-I) scores.

CONTACTS AND LOCATIONS:
Overall Officials: Karthikeyan Ganapathy, MD, Principal Investigator — Alberta Health Services/ Envision Mind Care
Locations (1):
- Envision Mind Care, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No